CLINICAL TRIAL: NCT04770714
Title: Comparison of Breast MRI Versus Contrast Enhanced Mammography Prior to Surgery in Breast Cancer Patients: a Randomized Controlled Trial
Brief Title: Prospective Comparison of Breast MRI vs Contrast Mammography Prior to Surgery in Breast Cancer Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No Participants enrolled.
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Michael Morris, Clinical Assistant Professor, Radiology, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010134480
Record Dates: First submitted 2021-01-19; First posted 2021-02-25 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Breast MRI (Other): Patients in this arm will be randomized to receive a Breast MRI in order to delineate the extent of a known cancer and / or assess for the presence of occult secondary cancers
  Interventions: Diagnostic Test: Breast MRI
- Contrast Enhanced Mammography (Other): Patients in this arm will be randomized to receive a Contrast Enhanced Mammograph in order to delineate the extent of a known cancer and / or assess for the presence of occult secondary cancers
  Interventions: Diagnostic Test: Contrast Enhanced Mammography

INTERVENTIONS:
Diagnostic Test: Breast MRI — Standard of Care Breast MRI
  Arms: Breast MRI
Diagnostic Test: Contrast Enhanced Mammography — Standard of Care Contrast Enhanced Mammography
  Arms: Contrast Enhanced Mammography

SUMMARY:
In current clinical practice, women with biopsy proven breast cancer can be sent for breast magnetic resonance imaging (MRI) or contrast enhanced mammography (CEM) prior to surgery in order to delineate the extent of a known cancer and / or assess for the presence of occult secondary cancers. This study seeks to compare the global costs (based on actual reimbursement rates) of CEM/breast MRI, downstream imaging testing, and diagnostic procedures in women randomized to breast MRI versus CEM. Secondary goals are to compare patient preferences for CEM vs MRI and clinically relevant outcomes (e.g. conversion from lumpectormy to mastecomy).

DETAILED DESCRIPTION:
This is a pilot randomized controlled trial comparing the global costs of two standard of care imaging techniques in patients with a new breast cancer diagnosis and planned breast conservation surgery. Patients enrolled in this study will be randomized to either CEM or breast MRI. The purpose of this study is to compare the global costs (based on actual reimbursement rates) of initial imaging modality (CEM or breast MRI), downstream imaging related to breast cancer evaluation, and diagnostic breast procedures in women randomized to breast MRI versus CEM.

Secondary endpoints include assessment of patient's reported satisfaction with the initial imaging technique received (CEM versus MRI), quantifying differences in health-related quality of life (as assessed by the patient reported Euro quality of life 5D questionnaire), rate of conversion from planned lumpectomy to mastectomy, and rate of re-operation for positive margins.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years or older with newly diagnosed breast cancer and planned breast conservation surgery
* Clinically indicated referral for breast MRI or contrast mammogram prior to surgery
* Provision of informed consent

Exclusion Criteria:

* Planned neoadjuvant chemotherapy
* Patients that are medically unstable
* Pregnancy
* Patients with known contraindication to contrast mammography, including:

  * Glomerular filtration rate <30
  * Known adverse reaction to iodinated contrast material
* Patients with known contraindication to Breast MRI including:

  * Glomerular filtration rate <30
  * Known adverse reaction to gadolinium contrast material
  * Non-MRI conditional device or catheter
  * Brain aneurysm clip implanted before 1995
  * Cochlear implant
  * Ocular foreign body (e.g. metal shavings)
  * Insulin pump
* Patients unable to read and understand English or Spanish (i.e. an inability to complete study questionnaires)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Global Costs | Through Study Completion (2 years)
  The Primary outcome is to compare the global costs (based on actual reimbursement rates) of initial imaging modality (CEM or breast MRI), downstream imaging related to breast cancer evaluation, and diagnostic breast procedures in women randomized to breast MRI versus CEM.

SECONDARY OUTCOMES:
Patient Satisfaction using modified Likert scale | Through Study Completion (2 years)
  Patient's reported satisfaction with the initial imaging technique received (CEM versus MRI) will be assessed via Post-Imaging questionnaires designed to gauge patient's opinions about the imaging technique they received.
Health-Related Quality of Life | Through Study Completion (2 years)
  quantifying differences in health-related quality of life (as assessed by the patient reported Euro quality of life 5D questionnaire)
Rate of Conversion | Through Study Completion (2 years)
  Rate of conversion from planned lumpectomy to mastectomy
Rate of Re-Operation | Through Study Completion (2 years)
  rate of re-operation for positive margins

CONTACTS AND LOCATIONS:
Locations (1):
- Banner University Medical Center Phoenixq, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
Study results will be shared on ClinicalTrials.gov in aggregate form.